CLINICAL TRIAL: NCT01206881
Title: A Phase II Study of Neoadjuvant Treatment With Pegylated Liposomal Doxorubicin (Caelyx) and Cyclophosphamide +/- Trastuzumab Followed by Docetaxel in Patients With Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Pegylated Liposomal Doxorubicin and Cyclophosphamide +/- Trastuzumab Followed by Docetaxel in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Malgorzata K. Tuxen, MD, phd, consultant, Department of Oncology, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO5903, EudraCT 2008-007951-29
Record Dates: First submitted 2010-09-13; First posted 2010-09-22 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant; liposomal doxorubicin; PET scan
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin — 35 mg/m2, IV, day 1 every 21 days, 4 cycles
  Other Names: cyclophosphamide, 4 cycles; docetaxel, 4 cycles; trastuzumab, 8 cycles

SUMMARY:
The purpose of this study is to determine the efficacy of neoadjuvant treatment with pegylated liposomal doxorubicin (Caelyx) and cyclophosphamide +/- trastuzumab followed by docetaxel in patients with locally advanced, inflammatory breast cancer or with a primary tumor > 5 cm.

DETAILED DESCRIPTION:
Patients with locally advanced or inflammatory breast cancer have a very bad prognosis. Several studies have shown that patients who receive a pathological complete response have the best prognosis. Neoadjuvant chemotherapy including anthracyclines and taxanes has become established as a standard option in the multidisciplinary management of this group of patients. In HER2 positive patients, chemotherapy in combination with trastuzumab is therapeutically attractive. Recent studies have also demonstrated that evaluation with PET-CT scan can be used to stratify treatment and monitor early response to neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven breast cancer
* inflammatory, locally advanced breast cancer or a tumor > 5 cm
* ECOG performance status < 2
* LVEF > 50% measured by MUGA (HER2 positive patients)
* adequate bone marrow, liver and renal function
* written informed consent must be obtained

Exclusion Criteria:

* another malignancy within 5 years prior to study entry
* concurrent treatment with an investigational agent
* other disease or condition that contraindicates participation in the study
* pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
clinical response rate | 24 weeks
  evaluation of treatment efficacy every 2.cycle

SECONDARY OUTCOMES:
pathological response rate, response rate as defined by PET-CT scan, mammography and ultrasound, evaluation of toxicity of the combination regimen | up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata K Tuxen, MD, Principal Investigator — Herlev Hospital, Department of Oncology; Ulla B Tange, MD, Principal Investigator — Rigshospitalet, Denmark; Soeren Cold, MD, Principal Investigator — Odense University Hospital; Susanne B Søndergaard, MD, Principal Investigator — Herlev Hospital; Henrik Petersen, MD, Principal Investigator — Odense University Hospital; Inger Hoejris, MD, Principal Investigator — Aarhus University Hospital; Anni Eskild-Jensen, MD, Principal Investigator — Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Tuxen MK, Cold S, Tange UB, Balslev E, Nielsen DL. Phase II study of neoadjuvant pegylated liposomal doxorubicin and cyclophosphamide +/- trastuzumab followed by docetaxel in locally advanced breast cancer. Acta Oncol. 2014 Oct;53(10):1440-5. doi: 10.3109/0284186X.2014.921727. Epub 2014 Jul 3. No abstract available. PMID 24991893